CLINICAL TRIAL: NCT02280915
Title: Assessment of the Bioavailability of Iron in Iron Fortified Savoury Food Product in Healthy Women
Brief Title: Bioavailability of Iron From Savoury Food Product
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Unilever R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: FDS-SAV-1615
Record Dates: First submitted 2014-10-21; First posted 2014-11-03 (Estimated); Last update posted 2015-05-01 (Estimated); Status verified 2015-04

CONDITIONS: Healthy; Iron Deficiency
Keywords: female; subjects
MeSH Terms: conditions — Iron Deficiencies

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Fortified savoury food product 1 (Experimental): Savoury food product fortified with iron
  Interventions: Other: Savoury food product
- Fortified savoury food product 2 (Experimental): Savoury food product fortified with iron
  Interventions: Other: Savoury food product
- Fortified savoury food product 3 (Experimental): Savoury food product fortified with iron
  Interventions: Other: Savoury food product
- Fortified savoury food product 4 (Experimental): Savoury food product fortified with iron
  Interventions: Other: Savoury food product

INTERVENTIONS:
Other: Savoury food product

SUMMARY:
The study is designed to assess the bioavailability of iron from 4 different iron fortified savoury food products

ELIGIBILITY:
Inclusion Criteria:

* Healthy female subjects;
* Age > 18 and < 40 years at screening;
* Body weight <65 kg;
* Apparently healthy: no medical conditions which might affect study measurements (judged by study physician);
* With iron deficiency (Serum ferritin <15µg/L);
* Currently not smoking and being a non-smoker for at least six months and no reported use of any nicotine containing products in the six months preceding the study and during the study itself;
* Willing and able to participate in the study; Having given a written informed consent.

Exclusion Criteria:

* Blood donation or significant blood loss over the past 6 months;
* Reported use of any medically- or self-prescribed diet;
* Use of medication (except oral contraceptives)
* Use of vitamin or mineral supplements and unwillingness to discontinue their use two weeks prior the study and during the study;
* Is pregnant or will be planning pregnancy during the study period;
* Is lactating or has been lactating in the 6 weeks before pre-study investigation and/or during the study period;
* Known gastrointestinal or metabolic disorders;
* Participation in another clinical trial during the last 30 days prior to the beginning of the study.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2014-10; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
To assess the absolute bioavailability of iron from 4 different iron fortified savoury food products | 15 days
  Amounts of Fe isotopic label present in the blood 14 days after administration of the fortified savoury food product will be calculated based on measured shifts in the iron isotope ratios in the blood samples (Day 15) compared to baseline and the amount of iron circulating in the body

SECONDARY OUTCOMES:
To assess the relative bioavailability of iron from iron fortified savoury food products | 15 days
  The absolute bioavailability results of each of the iron fortified savoury products as obtained under the primary objective will be compared with each other

CONTACTS AND LOCATIONS:
Overall Officials: Diego Moretti, Principal Investigator — ETH
Locations (1):
- Laboratory of human nutrition - ETH, Zurich, Switzerland